CLINICAL TRIAL: NCT03126656
Title: Effects of Testosterone on Myocardial Repolarization in Patients With Hypogonadism With/Without Chronic Heat Failure (NYHA Class I-II)
Brief Title: Effects of Testosterone on Myocardial Repolarization
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Gianfranco Piccirillo, Director Syncope Unit I Clinica Medica, Policlinico Umberto I, Rome, Italy, Clinical Professor, University of Roma La Sapienza
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TECHF001
Record Dates: First submitted 2017-04-19; First posted 2017-04-24 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Hypogonadism; Chronic Heart Failure
Keywords: testosterone; chronic heart failure
MeSH Terms: conditions — Hypogonadism | interventions — testosterone undecanoate

ARMS (3):
- Hypogonadic with chronic heart failure (Experimental): patients suffering from mild to moderate heart failure (LVEF ≥ 40%, NYHA I-II), and hypogonadism (plasma testosterone levels <11.4 nmol / L);
  Interventions: Drug: Testosterone Undecanoate
- Hypogonadic (Experimental): patients just with hypogonadism (testosterone <11.4 nmol / L) in the absence of documented cardiovascular disease
  Interventions: Drug: Testosterone Undecanoate
- chronic heart failure (No Intervention): patients suffering from mild to moderate heart failure (LVEF ≥ 40%, NYHA I-II) with normal testosterone levels(plasma testosterone levels > 11.4 nmol / L), in optimized standard therapy for heart failure

INTERVENTIONS:
Drug: Testosterone Undecanoate — just hypogonadic patients enrolled received hormone replacement therapy with testosterone undecanoate 1000 mg/4ml intramuscular (IM) at baseline, after 6 weeks and 12 weeks after the first evaluation
  Arms: Hypogonadic; Hypogonadic with chronic heart failure

SUMMARY:
The main of the study is to evaluate the effect of testosterone on ventricular repolarization in patients with mild heart failure, at risk for sudden cardiac death. The electrocardiographic markers studied are QT variability index, the short term variability index.

DETAILED DESCRIPTION:
Background:

It has been widely demonstrated in experimental cardiology that estrogen may play a protective role on cardiovascular system, reducing myocardial damage in ischemia-reperfusion injury. Poor are the contributions of the effects of estrogen in the presence of testosterone which also showed potentially cardioprotective effects. Recently it has emerged strong evidence showing that the increase in the repolarization phase of myocardial duration and its temporal dispersion are predictive markers of cardiac death in post-ischemic dilated cardiomyopathy. In addition, the temporal dispersion of the final part of the repolarization phase (Tpeak-Tend) is specifically predictive for sudden cardiac death. In fact, the investigators propose the following plan of experimental study. It will be measured by the duration of the repolarization phase and its basal temporal dispersion and the peak of the heart rate obtained during stress test, in male subjects before and during testosterone replacement therapy.

Patients evaluation baseline, after 1 month and after 6 months of follow up:

Endocrinological evaluation with measurement of body weight, height, BMI calculation and (digital rectal examination) DRE, blood sample.

Laboratory:

Dosage of serum total testosterone, total and free PSA, blood count.

Cardiological evaluation:

1. Patient's clinical objective examination: measurement of blood pressure and basal heart rate.
2. Traditional resting electrocardiogram 12-lead ECG in the supine position and 50 to 25 mm / sec, 10 millivolts.
3. Electrocardiographic single lead computerised registration (DI, D II and D III) of 5 minutes baseline and 5 minutes with controlled breathing (15 breaths / min), using the Spectralink 2011 program, which allows us to identify and calculate the variables object of this study;
4. Stress cycle electrocardiogram by modified Bruce protocol (25 watts every 2 minutes). The test is interrupted reaching 90% of the maximum heart rate, calculated based on the age of the patient, or to muscular exhaustion. A single lead electrocardiographic recording is started in the 10 minutes period after stress test, using Spectralink 2011 which allows investigators to calculate the variables studied.
5. trans thoracic echocardiogram with assessment of ejection fraction and any kinetic alterations in contractility and / or valvular heart disease, degree of possible diastolic dysfunction (E / A), size (interventricular septum, posterior wall, end-systolic and end-diastolic diameter in mm) and volumes (end-diastolic and end-systolic volume) of the left and right ventricle sections.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 70 aa with blood testosterone values <11.4 nmol / L;
* Sinus rhythm at 12-lead ECG;
* Hypogonadism: Total Testosterone <3.5 ng / ml or Free testosterone <250 pmol / L (10 pg / mL) detected (8: 00-11: 00 am) in two successive measurements taken baseline and confirmed at 7 days apart, reduced libido and / or at least two symptoms of hypogonadism evaluated AMS questionnaire
* previous myocardial infarction and relief echocardiographic fraction of left ventricular ejection greater than or equal to 40% (in chronic heart failure patients);
* stable clinical and hemodynamic conditions for more than three months;
* No therapeutic changes in the last 3 months;
* signing the informed consent.

Exclusion Criteria:

* therapy with testosterone undertaken within 6 months of enrollment or other therapy with steroids undertaken within 3 months thereafter
* Clinical history of prostate cancer
* elevated PSA values (adjusted for age)
* digital rectal exploration (DRE) suggestive of prostate cancer
* Symptoms of benign prostatic hypertrophy (BPH) with severe obstructive symptoms
* Hematocrit> 52% at baseline
* History of clinically significant hepatic, hematological, renal pathology
* Clinical history of breast cancer
* Hyperprolactinemia or other endocrine diseases (empty sella syndrome and pituitary expansive diseases measured by MRI)
* Age less than 40 or older than 70 years;
* Severe left ventricular systolic dysfunction (left ventricular ejection fraction <40%) and / or echocardiographic evidence of severe valvular disease;
* chronic atrial fibrillation or frequent extrasystoles (> 1 extrasystole / min);
* Presence of complete branch block;
* Unstable clinical and hemodynamic conditions and / or changes in therapy over the last three months;
* Presence of prostatic hyperplasia decisive severe obstruction to uroflow study;
* neoplasms diagnosed and treated less than five years later;
* Any other condition that medical judgment precludes patient safety

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — just male patients with hypogonadism or chronic heart failure or both are eligible
Enrollment: 123 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
QT duration reduction | baseline (before testosterone administration), after 1 month and after 6 months of follow up
  Reduction of the absolute QT interval value and its space and time dispersion

SECONDARY OUTCOMES:
hypogonadism treatment | baseline (before testosterone administration), after 1 month and after 6 months of follow up
  restoration of normal testosterone blood levels